CLINICAL TRIAL: NCT04134611
Title: Use of Hyaluronic Acid Injection After Arthroscopic Lateral Release in Patellar Compression Syndrome With Degenerative Cartilage Changes: Randomized Control Trial
Brief Title: Use of Hyaluronic Acid Injection in Lateral Patellar Compression With Femoral Condylar Degenerative Changes After Arthroscopic Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, Assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMU/Sherwan6
Record Dates: First submitted 2019-10-17; First posted 2019-10-22 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Anterior Knee Pain Syndrome
Keywords: Hyaluronic acid injection; Knee Arthroscopy; lateral patellar retinaculae.; lateral patellar compression syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee arthroscopy with Hyaluronic acid injection (Active Comparator): Those patients who received hyaluronic acid injection
  Interventions: Device: Hyaluronic acid injection
- Knee arthroscopy without Hyaluronic acid injection (Active Comparator): Knee arthroscopy who did not Hyaluronic acid injection
  Interventions: Device: No injection of Hyaluronic acid

INTERVENTIONS:
Device: Hyaluronic acid injection — Injection of Hyaluronic acid in knees of those who has degenerative changes after arthroscopic treatment of lateral patellar compression syndrome
  Arms: Knee arthroscopy with Hyaluronic acid injection
Device: No injection of Hyaluronic acid — No injection of Hyaluronic acid was done
  Arms: Knee arthroscopy without Hyaluronic acid injection

SUMMARY:
Ninety patients are involved in this study, who underwent arthroscopic lateral patellar release for lateral patellar compression syndrome and they had patellofemoral degenerative lesion, which diagnoses by MRI preoperatively and proved by arthroscopic examination to be early stages of degenerative changes with no loss of articular surface. The patients were divided in to two groups (A and B). Group A (45 patients) were treated by local injection of Hyaluronic acid intraarticularly, and Group B (45 patients) were no injection intraarticular.

DETAILED DESCRIPTION:
This study was done by one orthopedic surgeon in two hospitals. Ninety patients are involved in this study, who underwent arthroscopic lateral patellar release for lateral patellar compression syndrome and they had patellofemoral degenerative lesion, which diagnoses by MRI preoperatively and proved by arthroscopic examination to be early stages of degenerative changes with no loss of articular surface. The patients were divided in to two matched groups (A and B) regarding the age and gender; Group A (45 patients) were treated by local injection of Hyaluronic acid intraarticularly, 2 weeks after arthroscopy and were followed by VAS of knee pain for one year at (3) months, (6) months and (12) months, and Group B (45 patients) were no injection intraarticular. The study started on June (2017) and ends on March (2020). injection of Hyaluronic acid was used and followed in the same way. All patients presented with anterior knee pain which failed to respond to conservative treatment for 6 weeks or recurrent of symptoms after stopping of conservative treatment which involved changes of life style and NSAID. MRI done for all patients before operation.

ELIGIBILITY:
Inclusion Criteria:

* Lateral patellar compression syndrome

Exclusion Criteria:

* Patellar instability.
* Smoking.
* Diabetes Mellitus.
* Previous knee surgery.

Ages: 26 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Visual analogue score of knee pain | The VAS for knee pain was measured 24 months after operation
  Visual analogue score of knee pain describe knee pain from degree 0 where no pain to degree 10 where is severe pain
Kujala score | Preoperative assessment and 2 year postoperatively
  Kujala score questionnaire up to 100

CONTACTS AND LOCATIONS:
Locations (1):
- Sherwan Hamawandi, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Hamawandi SA. Use of hyaluronic acid injection after arthroscopic release in lateral patellar compression syndrome with degenerative cartilage changes: randomized control trial. BMC Musculoskelet Disord. 2021 Jan 6;22(1):24. doi: 10.1186/s12891-020-03876-0. PMID 33407337